

## CONSENT TO TAKE PART IN A RESEARCH STUDY

Title of Study: DBT Skills Video Intervention for Chinese and Chinese American College Students

Principal Investigator: Qingqing Yin, MS

**STUDY SUMMARY:** This consent form is part of an informed consent process for a research study, and it will provide information that will help you decide whether you want to take part in this study. It is your choice to take part or not.

The **purpose of the research** is to evaluate a brief coping skills video intervention delivered via smartphone. If you take part in the research, over the next 20 minutes you will be asked to complete some surveys that ask about your demographics and mental health. You will then be provided with instruction on how to download and use Catalyst By MetricWire (smartphone app) on your device. Over the next 4 weeks, you will be asked to complete a brief survey each day, on MetricWire, that will assess your emotional health. If you are placed into an intervention group, during 2 of these weeks you will also receive daily skills videos for 14 days that we will ask you to view and answer a few questions about. This is expected to take about 3-8 minutes per day to answer the surveys and watch the videos. Your total time in the study will be 4 weeks.

**Possible harms or burdens** of taking part in the study may be experiencing psychological distress while answering survey questions about your emotional health. Possible benefits of taking part may include learning ways to better cope with stressors. However, it is possible that you may not receive any direct benefit from taking part in this study.

An alternative to taking part in the research study is to choose to not take part in it.

The information in this consent form will provide more details about the research study to help you decide if you choose to take part in it. If you have any questions now or during the study, you should feel free to reach out to the study team and expect to be given answers you completely understand. After all your questions have been answered and you wish to take part in the research study, you will be asked to sign this consent form. You are not giving up any of your legal rights by agreeing to take part in this research or by signing this consent form.

## Who is conducting this study?

The Principal Investigator of this research study is Qingqing Yin, MS, who is a PhD student in clinical psychology at Rutgers University. Principal Investigator has the overall responsibility for the conduct of the research. However, there are often other individuals who are part of the research team.

Qingqing Yin may be reached at <a href="mailto:qy93@rutgers.edu">qy93@rutgers.edu</a>;732-630-8690; Psychology, 152 Frelinghuysen Rd, Rutgers University, Piscataway, NJ 08854.

#### Why is this study being done?

This study is being conducted to evaluate a coping skills intervention that is delivered remotely via short videos for college students who identify as Chinese or Chinese American. Despite pressing mental health needs, psychotherapy delivered in traditional format is unlikely to reach and benefit Chinese individuals



due to low treatment seeking and high dropout rates. These short videos may help provide coping skills for those who are interested in improving emotional health but not receiving mental health treatments.

## Who may take part in this study and who may not?

We are looking for undergraduate and graduate students to take part in this study who are at least 18 years of age, identify as Chinese or Chinese American, currently enrolled at Rutgers (on campus or remote), and are not currently receiving routine mental health services. We also want to enroll people who have an iOS or Android smartphone that is compatible with an research App, Catalyst by MetricWire (hereafter referred to as MetricWire). You may not be eligible for the study if you cannot speak or read English or if you are unable to provide written informed consent for any reason.

## Why have I been asked to take part in this study?

You have been invited to take part in this study because you completed a brief online screening that has identified you as an eligible participant.

### How long will the study take and how many subjects will take part?

We will enroll up to 150 participants to take part in this study. Should you choose to take part in this study, your participation will last for approximately 4 weeks.

## What will I be asked to do if I take part in this study?

If you choose to take part in this study, you will be randomized to one of three study groups, including one assessment-only group and two intervention groups that only differ in the sequence in which the skills videos are delivered. You will have a two-thirds chance of being assigned to an intervention group and a one-third chance of being placed in the assessment-only group.

Your participation in this study includes the following:

- Baseline Assessment: We will first ask you to complete a series of self-report surveys online
  that will include questions about your demographic information and mental health. We will then
  ask you to download the app, MetricWire, to your smartphone. Instructions on how to install and
  use the app will be provided. The baseline assessment will occur entirely online and take about
  20 minutes to complete.
- 2. Daily Smartphone Surveys: Over the next 4 weeks, we will ask you to complete up to a brief survey each day via MetricWire. You will be prompted to fill out these surveys by push notifications. These surveys will include questions about your emotional health such as your current emotion or use of coping skills. It is expected to take about 3 minutes each day to complete these surveys.
- 3. Coping Skills Videos: If you are placed into the intervention groups, you will also receive up to 14 brief coping skills videos via the smartphone app once per day for 2 weeks. This will occur approximately 1 week after you begin to complete the daily smartphone surveys. During this time, you will be asked to watch the video, practice the skill, and answer some questions about the video. There are two intervention groups that differ in the sequence in which the videos are delivered. This is expected to take about 5 minutes per day.

What are the risks of harm or discomforts I might experience if I take part in this study?

There are no risks of physical harm to taking part in this study. The risks of harm or discomforts associated with this study involve the possibility of experiencing distress while answering questions about your emotion health and daily stressors. However, you can skip any question that you feel uncomfortable with or do not wish to answer. Another potential risk involves potential breach of confidentiality or data security. We will take several measures to protect your confidentiality and data security as described

Protocol Version Date: Pro2023001220 Version 2.0 (August 2023)



below. We also encourage you to complete daily surveys promptly when notified to prevent your study participation from being seen by others in your environment.

## In case of high distress, please consider the following university resources:

- Rutgers Counseling, Alcohol and Other Drug Assistance Program & Psychiatric Services (CAPS); 848-932-7884; 17 Senior Street, New Brunswick, NJ 08901; Monday-Friday, 8:30am-4:30pm
- Rutgers University Police Department (RUPD); 848-932-7211
- Rutgers University Behavioral Health Care Acute Psychiatric Services (APS) Middlesex County; 855-515-5700

### Are there any benefits to me if I choose to take part in this study?

The potential benefits of taking part in this study include helping you better cope emotionally when faced with stressors. After the completion of the study period, all coping skills videos will be made available to you, regardless of whether you were placed into the intervention groups or not. However, it is possible that you may not receive any direct benefit from taking part in this study. Additionally, on a broader level, information from this study will be used to evaluate this innovative form of intervention among a culturally unique and diverse group thereby contributing to efforts to increase access to mental health resources.

## What are my alternatives if I do not want to take part in this study?

There are no alternative treatments available. Your alternative is to not take part in this study.

# How will I know if new information is learned that may affect whether I am willing to stay in the study?

During the study, you will be updated about any new information that may affect whether you are willing to continue taking part in the study. If new information is learned that may affect you after the study or your follow-up is completed, you will be contacted.

### Will I receive the results of the research?

In general, we will not give you any individual results from the study. However, if you are interested in reading the results of the study, you may contact the Principal Investigator who will email you the research article once published.

#### Will there be any cost to me to take part in this study?

There will not be any cost to you to take part in this study. The research App we will ask you to install on your phone requires very little data and can upload over Wi-Fi.

#### Will I be paid to take part in this study?

If you complete the baseline assessment and at least 20 out of 28 daily surveys over 4 weeks, you may choose to receive \$30 or 4 research participation units (RPUs) via the SONA/Human Subject Pool system for compensation. If you complete 25 or more surveys, you will receive an additional \$10 or an additional 1 RPU (i.e., total of \$40 or 5 RPUs). If you complete not as many as 20 surveys, but at least 7 daily surveys, you will receive \$10 or 1 RPU. You may choose to receive payment or RPUs only (not both), and the payment will be in the form of e-Gift-Cards sent via email.

#### How will information about me be kept private or confidential?

All efforts will be made to keep your personal information in your research record confidential, but total confidentiality cannot be guaranteed. Should you choose to participate in this study, information from the screener (e.g., email address, RUID) may be kept and used to contact you during the study. All data will be collected using secure software and App, and data collected will be recorded into secure electronic forms and transferred onto a password-protected cloud server. Research data will be linked with deidentified ID numbers, and no identifiable data will be stored alongside these data. Electronic consent



forms, not linked to participant ID numbers, will also be temporarily stored onto secure electronic forms and transferred onto the password-protected server. Access to the research data collected will be strictly restricted to the research team.

The research team may use or share your information collected or created for this study with the following people and institutions:

- Rutgers University investigators involved in the study
- The Rutgers University Institutional Review Board and Compliance Boards
- The Office for Human Research Protections in the U.S. Dept. of Health and Human Services

A description of this clinical trial will be available on <u>ClinicalTrials.gov</u>, as required by U.S. law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

## What will happen to my information collected for this research after the study is over?

After the study is over, information that could identify you will be removed, and de-identified data collected for this research may be used by investigators for other research without obtaining additional informed consent from you.

## What will happen if I do not wish to take part in the study or if I later decide not to stay in the study?

It is your choice whether to take part in the research. You may choose to take part/not to take part or you may change your mind and withdraw from the study at any time. If you do not want to enter the study or decide to stop taking part, your relationship with the study staff will not change, and you may do so without penalty and without loss of benefits to which you are otherwise entitled. Your decision to participate/withdraw will not be communicated to anyone outside of the research team.

You may also change your mind and not allow the continued use of your information at any time. If you take away your permission, your information will no longer be used or shared in the study. However, data that has already been used or shared with others cannot be withdrawn. If you change your mind later for use of your information in research, you must write to the Principle Investigator.

## Who can I contact if I have questions?

If you have questions, concerns or complaints about the research or if you feel you may have suffered a research related injury, you can contact the Principal Investigator, Qingqing Yin, MS, at: <a href="mailto:qy93@rutgers.edu">qy93@rutgers.edu</a>; 732-630-8690; Psychology, 152 Frelinghuysen Rd, Rutgers University, Piscataway, NJ 08854. You may also contact the faculty advisor, Shireen Rizvi, PhD, at: <a href="mailto:slrizvi@gsapp.rutgers.edu">slrizvi@gsapp.rutgers.edu</a>; 848-445-3942, Psychology, 152 Frelinghuysen Rd, Rutgers University, Piscataway, NJ 08854.

If you have questions, concerns, problems, information or input about the research or would like to know your rights as a research subject, you can contact the Rutgers IRB or the Rutgers Human Subjects Protection Program via phone at (973) 972-3608 or (732) 235-2866 or (732) 235-9806 OR via email irboffice@research.rutgers.edu, or you can write us at 335 George Street, Liberty Plaza Suite 3200, New Brunswick, NJ 08901

If you choose to participate in this study, you will automatically receive an electronic copy of this informed consent to your email. Please retain (print or save) a copy of this form for your records.

By selecting "I Agree" and providing your electronic signature you certify that you have read this entire consent form, understand the statements above, and will consent to participate in this study.



If you do not wish to participant in this study, select "I Do Not Agree".

- I Agree
- I Do Not Agree

By selecting "I Agree", providing your electronic signature in the signature box, and pressing the "next" button, you certify that you have read this entire consent form, understand the statements above, and will consent to participate in this study.

[Qualtrics signature box here]

[Finish button here]